CLINICAL TRIAL: NCT04247048
Title: A Kinetic Study of Lipoprotein in Humans for a Better Understanding of Lipoprotein(a) Metabolism Under PCSK9 Variations (Hu-La-u-P Study)
Brief Title: Kinetic Study of Lp(a) and PCSK9 in Humans
Acronym: HuLaUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Centre de Recherche en Nutrition Humaine Ouest (CRNH) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC18_0281
Record Dates: First submitted 2019-09-02; First posted 2020-01-29 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Cholesterol; Metabolic Disorder; Lipoproteinemia
MeSH Terms: conditions — Metabolic Diseases | interventions — Leucine

STUDY DESIGN:
Intervention Model Description: Kinetic study of lipoprotein metabolism with stable isotope tracers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Patients with no major LDL cholesterol abnormalities (patients eligible for LDL-apheresis, eg LDL-C> 200 mg / dL for secondary prevention and 300 mg / LDL-C) dl in primary prevention)) and a level of Lp (a) <50 mg / dl
  Interventions: Other: infusion of tracer [5,5,5-2H3] -L-leucine
- High-dose group (Experimental): Patients with no major LDL-cholesterol abnormalities (LDL-apheresis eligible patients, eg LDL-C> 200 mg / dL for secondary prevention and 300 mg / dl in primary prevention)) and a level of Lp (a)> 80 mg / dl
  Interventions: Other: infusion of tracer [5,5,5-2H3] -L-leucine

INTERVENTIONS:
Other: infusion of tracer [5,5,5-2H3] -L-leucine — A bolus of 6ml of [5,5,5-2H3] -L-leucine tracers will be performed followed by an infusion of 90 ml of [5,5,5-2H3] -L-leucine infused over 14 hours. This tracer participates in protein synthesis and especially in the synthesis of all apolipoproteins and PCSK9. Blood samples will be taken at T0, T2min, T5min, T10 minutes, T30 minutes and then every hour until 14 hours (a total of 240 ml of blood will be collected) to measure the stable tracer enrichment in the proteins of interest.

SUMMARY:
The aim is to study the relationship between lipoprotein(a) [Lp(a)] and PCSK9 (Proprotein Convertase Subtilisin/Kexin type 9) in humans with a kinetic study of lipoproteins in patients with dramatic increase of Lp(a) and controls.

DETAILED DESCRIPTION:
Elevated plasma levels of lipoprotein(a) [Lp(a)] are independently associated with an increased risk of cardiovascular diseases (CVD). Recently an unexpected and significant 15 to 30 % reduction of Lp(a) was reported with PCSK9 (Proprotein Convertase Subtilisin/Kexin type 9) inhibitors. The relation between Lp(a) and PCSK9 are unclear and debated.

Kinetic studies of lipoprotein are an important tool to decipher the complexity of apolipoprotein metabolism in human. The comparison of apoprotein(a) and PCSK9 kinetic parameters of patients with extreme lipid disorder link to PCSK9 and apo(a) will allow to better understand the impact of PCSK9 on apo(a). From one previous in vitro study, the hypothesize is that PCSK9 increases the production rate and the assembly of Lp(a).

The objectives are to explore the relationship between the plasma concentration of PCSK9 and apo(a) production rate as well as the impact on the catabolic rate. Patients with extreme Lp(a) levels and healthy controls will be explored by performing a continuous infusion of deuterated leucine for 14 hours. LC/MS-MS will be used to analyze the samples and kinetic data of apo(a) and PCSK9 will be generated from a compartmental model. Tracer enrichment analysis could be complicated for proteins with low plasma concentrations as PCSK9. This issue will be solved with SPE and/or immune affinity concentration techniques. Non-parametrical test and multivariate analysis will be use to describe the relationship between these two variables.

This study will provide new knowledge on Lp(a) and PCSK9 metabolism and their interactions in humans.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 75 years
* For subjects in the "Control" group: Patients with no major LDL-cholesterol deficiency (patients eligible for LDL-apheresis, eg LDL-C> 200 mg / dL for secondary prevention and 300 mg / dl in primary prevention)) and a level of Lp (a) <50 mg / dl or
* For subjects in the "high-dose" group: Patients with no major LDL-cholesterol abnormalities (LDL-apheresis eligible patients, eg LDL-C> 200 mg / dL for secondary prevention and 300 mg / dl in primary prevention)) and a level of Lp (a)> 80 mg / dl Whenever possible, groups will be balanced for age, sex, familial forms of hypercholesterolemia and their major groups of mutations.

Exclusion Criteria:

* Patients treated with PCSK9 antibodies.
* Patients with acute illness and considered incompatible by the investigator
* Uncontrolled diabetes (HbA1c> 8.5%)
* Severe hepatic insufficiency
* Creatinine clearance <30 ml / min
* Patients not covered by a social security scheme or beneficiary of such a scheme
* Patients unable to understand and / or sign consent
* Pregnant or lactating women
* Minors
* Majors under guardianship or trusteeship or safeguard of justice

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
To study in humans by a study of the kinetics of apo (a), the relationships between the metabolism of Lp (a) and the plasma levels of PCSK9. | 14 hours after leucine infusion
  1. Correlation between PCSK9 plasma levels and apo (a) production rate (fractional production rate (RPF) and absolute production rate (APR)) in patients with Lp (a)> 80 mg / dl and control subjects with Lp (a) levels <30mg / dl.
  2. Correlation between PCSK9 plasma levels and apo (a) fractional clearance rate (FCR) in patients with Lp (a)> 80 mg / dl and control subjects with Lp (a) levels <30mg / dl.

SECONDARY OUTCOMES:
To evaluate the impact of PCSK9 metabolism on metabolic parameters of Lp (a). | 14 hours after leucine infusion
  Correlation between the PCSK9 (fractional production rate (RPF) and absolute production rate (APR) synthesis rate and the rate of synthesis and degradation of apo (a) (fractional production rate (FPR) and absolute production rate ( APR)) and fractional clearance rate (FCR) in patients with Lp (a)> 80 mg / dl and control subjects with Lp (a) <30mg / dl.
To evaluate the impact of PCSK9 metabolism on metabolic parameters of Lp | 14 hours after leucine infusion
  Correlation between PCSK9 (fractional clearance rate (FCR)) and the rate of synthesis and degradation of apo (fractional production rate (RPF) and absolute production rate (APR)) and (fractional clearance rate spleen (FCR)) in patients with Lp (a)> 80 mg / dl and control subjects with Lp (a) <30mg / dl.
To measure the impact of PCSK9 metabolism on metabolic parameters of Lp | 14 hours after leucine infusion
  Correlation between the production and degradation rates of Lp (a), PCSK9 and apoB100 in patients with Lp (a)> 80 mg / dl and control subjects with Lp (a) ) <30 mg / dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France